CLINICAL TRIAL: NCT07125534
Title: Alcohol and the Social Brain: An Alcohol-Administration Hyperscanning Study Employing a Within-Subject Design
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Catharine Fairbairn, Ph.D., University of Illinois at Urbana-Champaign
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2R01AA025969-01 (NIH)
Record Dates: First submitted 2025-08-09; First posted 2025-08-15 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Alcohol Drinking; Alcohol Use Disorder (AUD); Alcohol Intoxication; Alcohol; Harmful Use; Alcoholism; Binge Drinking
MeSH Terms: conditions — Alcohol Drinking; Alcoholism; Alcoholic Intoxication; Binge Drinking | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alcohol beverage administration (Experimental)
  Interventions: Drug: Alcohol beverage
- Control condition - non alcoholic beverage (Other)
  Interventions: Other: Control - non alcoholic beverage

INTERVENTIONS:
Drug: Alcohol beverage — This intervention involves the administration of an alcohol beverage (vodka mixed with juice or soda) in a controlled laboratory setting, targeting a blood alcohol concentration (BAC) of 0.08%. The alcohol is consumed over a 36-minute period in three equal parts.
  Arms: Alcohol beverage administration
Other: Control - non alcoholic beverage — This intervention involves the administration of a non-alcoholic control beverage in a controlled laboratory setting. The beverage is matched in volume and palatability to the alcohol condition but co
  Arms: Control condition - non alcoholic beverage

SUMMARY:
The study investigates the effects of alcohol consumption on social and individual behaviors using a within-subject design. Participants, aged 21-30, will attend two laboratory sessions approximately one week apart, participating as part of a dyad (pair). During one session, they will consume an alcoholic beverage, while in the other, they will receive a control beverage, with the order of conditions randomized. This design facilitates direct within-participant comparisons of behaviors and neural activity in intoxicated versus sober states.

To achieve these aims, the study employs EEG technology to explore intra-brain and inter-brain dynamics during social interactions. Additionally, validated self-report questionnaires will capture data on mood, social bonding, and other psychological variables. The findings are expected to enhance understanding of alcohol's role in social reward processes and contribute to developing evidence-based prevention and intervention strategies for alcohol use disorder.

DETAILED DESCRIPTION:
Objective:

Alcohol's ability to enhance social bonding and modulate mood in social contexts has been identified as a key factor contributing to its reinforcing properties and risk for Alcohol Use Disorder (AUD). While prior research has demonstrated alcohol's role in enhancing social interactions, laboratory studies often fail to replicate the real-world context in which most alcohol consumption occurs-social settings with familiar companions. This discrepancy limits our understanding of the mechanisms through which alcohol exerts its effects in social contexts.

This study is the first to employ EEG hyperscanning methods to investigate the inter- and intra-brain mechanisms underlying alcohol's social rewards within dyadic interactions. Specifically, the study aims to characterize how alcohol modulates social bonding, emotional regulation, and neural synchrony during social interactions, and to identify the cognitive and affective processes driving alcohol's reinforcing properties. The findings are expected to deepen understanding of the role of alcohol in social dynamics and inform interventions for AUD.

Study Population:

The study will recruit 200 participants, aged 21-30, who self-identify as regular social drinkers and with no reported history of severe alcohol use disorder.

Design:

This within-subject laboratory study involves two experimental sessions spaced approximately one week apart. Each session includes participants interacting in dyads with a stranger, where they will consume either a moderate dose of alcohol (target BAC ~0.08%) or a non-alcoholic control beverage, with the order randomized between sessions. Participants will engage in structured and unstructured tasks during each session, allowing for the evaluation of behavioral, emotional, and neural outcomes in both intoxicated and sober states.

* EEG Hyperscanning: Neural activity will be recorded simultaneously from both members of the dyad using EEG hyperscanning technology. This allows for the investigation of intra-brain processes (e.g., cognitive and emotional regulation) and inter-brain synchrony (e.g., neural alignment during social interactions).
* Tasks and Measures: Participants will complete tasks designed to assess social bonding, emotional regulation, and cognitive processing. Tasks include structured paradigms (e.g., music perception tasks and flanker task) and naturalistic social interactions. These are complemented by self-report measures assessing mood, social closeness, and perceptions of the interaction.
* Randomization and Counterbalancing: The order of alcohol versus control sessions will be randomized across participants to control for carryover effects.

Outcome Measures:

1. Neurophysiological Outcomes:

   Intra and Inter Brain Coupling (IBC):
   * Intra brain synchrony (within-subject): Coherence or phase-locking between brain regions within the same participant, compared across sober versus intoxicated states.
   * Inter brain synchrony (between-subject): Synchronization metrics (e.g., inter subject PLV, inter subject correlation) between paired participants, assessed separately in sober and intoxicated conditions

   Event Related Potentials (ERP):

   • Amplitudes and latencies of task-related ERP components, specifically Feedback Related Negativity (FRN), measured both for the operating ("player") and observing ("observer") participant, with comparisons across sobriety conditions
2. Behavioral and Psychological Outcomes:

   Self-reported mood and social bonding assessed pre- and post-interaction using validated measures such as the Inclusion of Other in Self Scale and the Biphasic Alcohol Effects Scale.

   Observational coding of nonverbal behaviors (e.g., facial expressions, body language) during dyadic interactions.
3. Drinking Behavior:

Longitudinal self-reports of drinking patterns and alcohol-related outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 21 and 30
* Regularly consumes alcohol

Exclusion Criteria:

* History of adverse reaction to the amount of beverage employed in the study
* Have a history of major problems associated with alcohol
* Take medications that could adversely interact with alcohol
* Have medical conditions that contraindicate alcohol administration
* Individuals with a history of skull fractures or who indicate discomfort with EEG procedures used
* Female participant is pregnant or trying to become pregnant

Ages: 21 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-08-09 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Inter-brain entrainment | During active laboratory beverage manipulation exposure (during or immediately after beverage administration, at which time participants in the alcohol condition will register a positive BAC)
  Synchronization metrics (e.g., inter-subject PLV, inter-subject correlation) between paired participants, assessed separately in sober and intoxicated conditions
Intra-brain entrainment | During active laboratory beverage manipulation exposure (during or immediately after beverage administration, at which time participants in the alcohol condition will register a positive BAC)
  The comparison of EEG signal synchronization within the same participant across the alcohol and non-alcohol conditions, reflecting intra-brain activity changes due to alcohol consumption during the hyperscanning task.
Event-Related Potentials (ERP) | During active laboratory beverage manipulation exposure (during or immediately after beverage administration, at which time participants in the alcohol condition will register a positive BAC)
  Feedback-Related Negativity (FRN), measured both for the operating ("player") and observing ("observer") participant, with comparisons across sobriety conditions
Ambulatory Drinking | 14 days
  Drinking behavior assessed outside the laboratory using ambulatory assessment
Longitudinal Drinking Problems | Up to 24 months post-baseline
  Drinking assessed at longitudinal follow-up

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Illinois at Urbana Champaign, Champaign, Illinois
  - University of Illinois Urbana-Champaign, Champaign, Illinois

IPD SHARING:
Plan to Share IPD: Yes
Data is being shared on the National Institute of Mental Health Data Archive